CLINICAL TRIAL: NCT00642070
Title: Host Response to Urinary Tract Infection in Women
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ann Stapleton, Professor, University of Washington
Other Study IDs: 31467-D; NIDDK 1 P50 AR049475-06;; 06-4836-D (Other: University of Washington Human Subjects Division)
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Urinary Tract Infection
Keywords: Current symptoms of urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood,serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Host: Women with current symptoms of a urinary tract infection

SUMMARY:
This study is being done to identify those elements of the immune response that may predispose a woman to recurrent urinary tract infection. We suspect that lesser effectiveness of certain components of the host response will lead to recurrent urinary tract infection. We will also evaluate the role that the bladder reservoir may play in recurrent urinary tract infection.

DETAILED DESCRIPTION:
Procedures subjects will undergo once they have read and signed the consent are:

Questions about their medical and sexual history and current symptoms of urinary tract infection. They will be asked to provide a clean catch urine sample. We will collect periurethral, vaginal and rectal swabs. Blood will collected. They will be given a diary to take home and record all episodes of sexual intercourse, contraceptive use, vaginal and urinary symptoms and medication use.

They will be given standard treatment for the current urinary tract infection. Follow-up visits will be scheduled 2 weeks,one month,two month and three month after initial visit.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-49 years
* Able to provide written informed consent
* diagnosis of acute cystitis with symptoms for fewer than 7 days

Exclusion Criteria:

* Not pregnant or planning pregnancy in next 3 months
* No chronic illness requiring medical supervision (e.g. diabetes mellitus)
* No known anatomic or functional abnormalities of the urinary tract
* No signs or symptoms suggestive of pyelonephritis (flank pain or tenderness, temperature over 100 degrees F, nausea or vomiting)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women between the ages of 18-49 with symptoms of a urinary tract infection for fewer than 7 days
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2008-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Determine elements of the immune response that may predispose a woman to recurrent urinary tract infection | 2017

CONTACTS AND LOCATIONS:
Overall Officials: Ann E Stapleton, M.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington/Hall Health Primary Care Center, Seattle, Washington, United States